CLINICAL TRIAL: NCT04063189
Title: A Prospective, Multicenter, Single Arm, Phase II Clinical Trial of Clarithromycin, Lenalidomide and Dexamethasone (BiRd Regimen) in the Treatment of the First Relapsed Multiple Myeloma
Brief Title: Clinical Trial of Clarithromycin, Lenalidomide and Dexamethasone in the Treatment of the First Relapsed Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, FengYan Jin, MD, PHD, Physician in Charge of Hematology Department, The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BiRd 2017-288-1
Record Dates: First submitted 2018-01-17; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Multiple Myeloma in Relapse
Keywords: Clarithromycin Lenalidomide Dexamethasone Regimen; Treatment Response; Survival
MeSH Terms: interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- First Relapsed Multiple Myeloma (Experimental)
  Interventions: Drug: Clarithromycin Lenalidomide Dexamethasone (BiRd) Regimen

INTERVENTIONS:
Drug: Clarithromycin Lenalidomide Dexamethasone (BiRd) Regimen — Clarithromycin 500mg，po，bid，d1-21; Lenalidomide 25mg，po，daily，d1-21 (dose according to creatinine clearance rate); Dexamethasone 20mg，po，daily，d1-2, 8-9,15-16, 22-23

SUMMARY:
BiRd regimen consisting of clarithromycin and Rd is safe and effective in NDMM. It can significantly increase ORR (up to 90.3%) , relief depth (≥VGPR), and prolong PFS to 43 months. In our previous study, thirty RRMM patients treated with BiRd regimen in 6 centers in China benefited.It suggested that BiRd regimen may not only improve overall efficacy of RRMM , especially long-term benefits, but also reverse Rd resistance in patients who fail to achieve any remission after multiline therapy.The study is a Prospective, Multicenter, Single Arm, Phase II Clinical Trial, which intend to recruit first relapse MM patients over 18 years old. Once included, patients will receive the treatment of Clarithromycin Lenalidomide Dexamethasone (BiRd) Regimen. (Clarithromycin 500mg，po，bid，d1-21; Lenalidomide 25mg，po，daily，d1-21 (dose according to creatinine clearance rate); Dexamethasone 20mg，po，daily，d1-2, 8-9,15-16, 22-23) And we will evaluate efficacy and adverse events of the BiRd regimen at a point of time predetermined.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed as symptomatic multiple myeloma.
2. the first relapse/progression with thalidomide, bortezomib or lenalidomide based current first-line treatment or resistance to the first-line treatment (previous treatment line number =1).
3. there must be measurable lesions to determine disease progression (PD): according to the IMWG 2016 efficacy evaluation criteria.
4. the expected survival time is longer than 3 months.
5. ECOG score less than 2 points.
6. the serum AST/ALT level <3 times higher than the normal value; the serum total bilirubin level<2 times of the normal value; creatinine clearance rate was ≥30ml/mi.
7. neutrophil count >1000/mm3 ; platelet count >75000/mm3 (if bone marrow plasma cell <50%) or >30000/mm3 (if the plasma cells in the bone marrow is not less than 50%).
8. women of childbearing age were negative for pregnancy before admission, and agreed to carry out pregnancy screening during the study (once a month until 4 weeks after the last dose), and agreed to use contraceptive measures within 3 months after the study and the last dose.
9. all patients were required to sign informed consent.

Exclusion Criteria:

1. under the age of 18
2. ECOG score >2
3. non secretory myeloma, defined as serum protein M < 1g/dL, urinary M protein < 200mg/24h and sFLCR ≤100mg/L
4. there is growing demand, pregnant or lactating women within one year
5. HIV infection
6. activity of HBV or HCV infection
7. 4 weeks before entering the group of thromboembolic events
8. not signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-21 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Every 2 months until disease progression or study completion，an average of 2 year
  According to the criteria of IMWG 2016

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by NCI-CTCAE v4.03 | Through study completion,an average of 2 year
  According to NCI-CTCAE version 4.03
Progression-Free Survival (PFS) | Through study completion, an average of 2 year
  PFS were calculated from the enrollment to the first instance of disease progression, relapse, or death
Overall Survival (OS) | Through study completion, an average of 2 year
  OS were calculated from the time of enrollment to death or the last follow-up
Duration of Response (DOR) | Through study completion, an average of 2 year
  the time from the first assessment of CR (complete response) or PR (partial response) to the first PD (Progressive Disease) or any cause of death

OTHER OUTCOMES:
Health-Related Quality of Life (HRQoL) | Every 6 months until disease progression or study completion，an average of 2 year
  According to the data of SF-36 Quality of Life Questionnaire Survey

CONTACTS AND LOCATIONS:
Overall Officials: Fengyan Jin, professor, Study Director — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Palumbo A, Anderson K. Multiple myeloma. N Engl J Med. 2011 Mar 17;364(11):1046-60. doi: 10.1056/NEJMra1011442. No abstract available. PMID 21410373
- [Background] Agarwal A, Chow E, Bhutani M, Voorhees PM, Friend R, Usmani SZ. Practical Considerations in Managing Relapsed Multiple Myeloma. Clin Lymphoma Myeloma Leuk. 2017 Feb;17(2):69-77. doi: 10.1016/j.clml.2016.11.010. Epub 2016 Nov 23. PMID 27986429
- [Background] Plesner T, Arkenau HT, Gimsing P, Krejcik J, Lemech C, Minnema MC, Lassen U, Laubach JP, Palumbo A, Lisby S, Basse L, Wang J, Sasser AK, Guckert ME, de Boer C, Khokhar NZ, Yeh H, Clemens PL, Ahmadi T, Lokhorst HM, Richardson PG. Phase 1/2 study of daratumumab, lenalidomide, and dexamethasone for relapsed multiple myeloma. Blood. 2016 Oct 6;128(14):1821-1828. doi: 10.1182/blood-2016-07-726729. Epub 2016 Aug 16. PMID 27531679
- [Background] Popat R, Brown SR, Flanagan L, Hall A, Gregory W, Kishore B, Streetly M, Oakervee H, Yong K, Cook G, Low E, Cavenagh J; Myeloma UK Early Phase Clinical Trial Network. Bortezomib, thalidomide, dexamethasone, and panobinostat for patients with relapsed multiple myeloma (MUK-six): a multicentre, open-label, phase 1/2 trial. Lancet Haematol. 2016 Dec;3(12):e572-e580. doi: 10.1016/S2352-3026(16)30165-X. Epub 2016 Nov 12. PMID 27843120
- [Background] Weber DM, Chen C, Niesvizky R, Wang M, Belch A, Stadtmauer EA, Siegel D, Borrello I, Rajkumar SV, Chanan-Khan AA, Lonial S, Yu Z, Patin J, Olesnyckyj M, Zeldis JB, Knight RD; Multiple Myeloma (009) Study Investigators. Lenalidomide plus dexamethasone for relapsed multiple myeloma in North America. N Engl J Med. 2007 Nov 22;357(21):2133-42. doi: 10.1056/NEJMoa070596. PMID 18032763
- [Background] Dimopoulos M, Spencer A, Attal M, Prince HM, Harousseau JL, Dmoszynska A, San Miguel J, Hellmann A, Facon T, Foa R, Corso A, Masliak Z, Olesnyckyj M, Yu Z, Patin J, Zeldis JB, Knight RD; Multiple Myeloma (010) Study Investigators. Lenalidomide plus dexamethasone for relapsed or refractory multiple myeloma. N Engl J Med. 2007 Nov 22;357(21):2123-32. doi: 10.1056/NEJMoa070594. PMID 18032762
- [Background] Hou J, Du X, Jin J, Cai Z, Chen F, Zhou DB, Yu L, Ke X, Li X, Wu D, Meng F, Ai H, Zhang J, Wortman-Vayn H, Chen N, Mei J, Wang J. A multicenter, open-label, phase 2 study of lenalidomide plus low-dose dexamethasone in Chinese patients with relapsed/refractory multiple myeloma: the MM-021 trial. J Hematol Oncol. 2013 Jun 19;6:41. doi: 10.1186/1756-8722-6-41. PMID 23782711
- [Background] Dimopoulos MA, Chen C, Spencer A, Niesvizky R, Attal M, Stadtmauer EA, Petrucci MT, Yu Z, Olesnyckyj M, Zeldis JB, Knight RD, Weber DM. Long-term follow-up on overall survival from the MM-009 and MM-010 phase III trials of lenalidomide plus dexamethasone in patients with relapsed or refractory multiple myeloma. Leukemia. 2009 Nov;23(11):2147-52. doi: 10.1038/leu.2009.147. Epub 2009 Jul 23. PMID 19626046
- [Background] Rossi A, Mark T, Jayabalan D, Christos P, Zafar F, Pekle K, Pearse R, Chen-Kiang S, Coleman M, Niesvizky R. BiRd (clarithromycin, lenalidomide, dexamethasone): an update on long-term lenalidomide therapy in previously untreated patients with multiple myeloma. Blood. 2013 Mar 14;121(11):1982-5. doi: 10.1182/blood-2012-08-448563. Epub 2013 Jan 8. PMID 23299315
- [Background] Niesvizky R, Jayabalan DS, Christos PJ, Furst JR, Naib T, Ely S, Jalbrzikowski J, Pearse RN, Zafar F, Pekle K, Larow A, Lent R, Mark T, Cho HJ, Shore T, Tepler J, Harpel J, Schuster MW, Mathew S, Leonard JP, Mazumdar M, Chen-Kiang S, Coleman M. BiRD (Biaxin [clarithromycin]/Revlimid [lenalidomide]/dexamethasone) combination therapy results in high complete- and overall-response rates in treatment-naive symptomatic multiple myeloma. Blood. 2008 Feb 1;111(3):1101-9. doi: 10.1182/blood-2007-05-090258. Epub 2007 Nov 7. PMID 17989313
- [Background] Kato H, Onishi Y, Okitsu Y, Katsuoka Y, Fujiwara T, Fukuhara N, Ishizawa K, Takagawa M, Harigae H. Addition of clarithromycin to lenalidomide/low-dose dexamethasone was effective in a case of relapsed myeloma after long-term use of lenalidomide. Ann Hematol. 2013 Dec;92(12):1711-2. doi: 10.1007/s00277-013-1761-x. Epub 2013 Apr 28. No abstract available. PMID 23625297
- [Background] Ghosh N, Tucker N, Zahurak M, Wozney J, Borrello I, Huff CA. Clarithromycin overcomes resistance to lenalidomide and dexamethasone in multiple myeloma. Am J Hematol. 2014 Aug;89(8):E116-20. doi: 10.1002/ajh.23733. Epub 2014 Apr 26. PMID 24723438